CLINICAL TRIAL: NCT00343226
Title: An Open, Randomized Pilot Study to Evaluate the Use of Basiliximab With an Optimized Cyclosporine Dosing on Renal Function in "de Novo" Liver Transplantation.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Novartis, Novartis
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CCHI621ABE02
Record Dates: First submitted 2006-05-30; First posted 2006-06-22 (Estimated); Last update posted 2010-08-25 (Estimated); Status verified 2010-08

CONDITIONS: Liver Transplantation
Keywords: Basiliximab, transplantation, liver, renal function
MeSH Terms: interventions — Basiliximab

INTERVENTIONS:
Drug: Basiliximab

SUMMARY:
The objectives of the study are:To compare the renal function of a quadruple immunosuppressive regimen (including basiliximab in combination with an optimized cyclosporine dose during the first weeks post-transplantation, mycophenolate mofetil and corticosteroids) versus a standard triple therapy regimen (including cyclosporine standard dose, mycophenolate mofetil and corticosteroids)

ELIGIBILITY:
Inclusion Criteria

* First cadaveric liver transplant
* ABO identical or compatible graft

Exclusion Criteria

* Multiple organ transplant
* renal impairment defined as glomerular filtration rate (GFR) < 30 ml/min
* Fulminant liver failure

Other protocol-defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2002-05; Primary Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Renal function (i.e. glomerular filtration rate) at 12 months post-transplantation

SECONDARY OUTCOMES:
Frequency and severity of rejection episodes before 6 and 12 months post-transplantation
Frequency of death, graft loss or retransplantation before 6 and 12 months post-transplantation
Adverse events
Duration of initial hospitalization and number or hospital re-admissions.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis, Study Director — Novartis